CLINICAL TRIAL: NCT03344042
Title: Effect of Epidural Opioid Administered in the First A Period on the Progress of Labour
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Jan Biławicz, Principal Investigator, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KB/46/2016
Record Dates: First submitted 2017-08-16; First posted 2017-11-17 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Anesthesia, Epidural; Opioid; Labor Pain
MeSH Terms: conditions — Labor Pain | interventions — Fentanyl; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant not aware of opioid administered
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fentanyl (Active Comparator): 100mcg Fentanyl administered into epidural space during regular contractions before cervical dilation
  Interventions: Drug: Fentanyl
- Sufentanyl (Active Comparator): 10mcg sufentanyl administered into the epidural space during regular contractions before cervical dilation
  Interventions: Drug: Sufentanil
- Control (No Intervention): No epidural analgesia

INTERVENTIONS:
Drug: Fentanyl — 100mcg Fentanyl
  Arms: Fentanyl
Drug: Sufentanil — 10mcg sufentanil
  Arms: Sufentanyl

SUMMARY:
Epidural anesthesia is used to relieve labour pain which helps reduce labour stress, increase comfort and improve cooperation with medical personnel. Administering opioid into the epidural space before cervical dilation of 4cm in the primigravida or 3cm in the multiparous can effectively reduce the pain levels with no effect on the labour progress. The aim of the study is to compare different opioids administered in this early labour stage.

ELIGIBILITY:
Inclusion Criteria:

* parturient in labour without cervical dilation and regular uterine contractions

Exclusion Criteria:

* no consent
* known allergy to administered opioid
* contraindications to epidural analgesia
* coagulopathies including platelet count of less than 100,000
* spine surgery in past

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-12-20 (Estimated); Study Completion 2018-12-20 (Estimated)

PRIMARY OUTCOMES:
Pain intensity according to Numerical Rating Scale (NRS) | up to 24 hours
  till 4cm cervical dilation in primigravida or 3cm multiparous

SECONDARY OUTCOMES:
Fetal heart rate | up to 24 hours
  till 4cm cervical dilation in primigravida or 3cm multiparous
Blood pressure parturient | up to 24 hours
  till 4cm cervical dilation in primigravida or 3cm multiparous
Heart rate of parturient | up to 24 hours
  till 4cm cervical dilation in primigravida or 3cm multiparous

CONTACTS AND LOCATIONS:
Locations (1):
- Uniwersyteckie Centrum Zdrowia Kobiety i Noworodka, WUM, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided